CLINICAL TRIAL: NCT01931527
Title: Effect of Plasma Uric Acid on Insulin Sensitivity, Endothelial Function and Inflammation
Brief Title: Effect of Reducing Uric Acid on Insulin Sensitivity and Oxidative Status
Acronym: UA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 06-0509 / 201104189
Record Dates: First submitted 2013-08-23; First posted 2013-08-29 (Estimated); Results first posted 2015-05-15 (Estimated); Last update posted 2018-08-14 (Actual); Status verified 2018-07

CONDITIONS: Obesity; Metabolic Syndrome; Hyperuricemia
Keywords: Obesity; Metabolic syndrome; Hyperuricemia
MeSH Terms: conditions — Obesity; Metabolic Syndrome; Hyperuricemia | interventions — rasburicase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Obese subjects with normal uric acid (No Intervention): Subjects with a body mass index = or > 30 kg/m² with normal uric acid (= or < 5 mg/dL)
- Obese subjects with high uric acid (Experimental): Subjects with a body mass index = or > 30 kg/m² with high uric acid (>6 mg/dL)
  Intervention: one single infusion of rasburicase (0.19 mg/kg FFM) infused over 30 min
  Interventions: Drug: Rasburicase

INTERVENTIONS:
Drug: Rasburicase — one single infusion of rasburicase (0.19 mg/kg FFM) infused over 30 min
  Other Names: Elitek
  Arms: Obese subjects with high uric acid

SUMMARY:
The purpose of this study is to learn more about what is the effect of uric acid on oxidative stress and on the way the body metabolizes sugar in obese people. Understanding this may lead to better diseases such as diabetes.

DETAILED DESCRIPTION:
It has been hypothesized that oxidative stress is involved in the pathogenesis of insulin resistance associated with obesity. Circulating uric acid (UA) is the body's major endogenous plasma antioxidant. Therefore, the investigators evaluated whether alterations in serum UA concentration affect: 1) systemic and skeletal muscle oxidative stress, 2) total antioxidant capacity, and 4) skeletal muscle insulin sensitivity during a hyperinsulinemic-euglycemic clamp.

ELIGIBILITY:
Inclusion Criteria:

* obese (BMI 30-45 kg/m²);
* serum UA concentration either ≥5 mg/dL or ≤4.0 mg/dL (297 µmol/L)],

Exclusion Criteria:

* renal dysfunction (serum creatinine >1.5 mg/dL);
* pregnancy or lactating;
* take urate-lowering agents, thiazide diuretics, prednisone or medications containing aspirin or other salicylates;
* history of xanthinuria, type 2 diabetes or other significant organ system dysfunction;
* have G6PD deficiency;
* use hormone-replacement or oral-contraceptive therapy;
* smoke tobacco;
* anemic (Hb <10 g/dl)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2006-07; Primary Completion 2008-06 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Klein, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Obese Subjects With Normal Uric Acid: Subjects with a body mass index = or > 30 kg/m2 with normal uric acid (= or < 5 mg/dL)
- Obese Subjects With High Uric Acid: Subjects with a body mass index = or > 30 kg/m2 with high uric acid (>6 mg/dL)
  Intervention: one single infusion of rasburicase (0.19 mg/kg FFM) infused over 30 min
  Rasburicase: one single infusion of rasburicase (0.19 mg/kg FFM) infused over 30 min
Period: Overall Study
Arm/Group | Obese Subjects With Normal Uric Acid | Obese Subjects With High Uric Acid
Started | 16 | 15
Completed | 16 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Obese subjects with low uric acid (<5mg/dL)
Groups:
- Low Uric Acid: 16 obese subjects (BMI 37.1±0.7 kg/m2) with uric acid <5mg/dL
- High Uric Acid: 15 obese subjects (BMI 37.1±0.7 kg/m2) with uric acid >6mg/dL
- Total: Total of all reporting groups
Arm/Group | Low Uric Acid | High Uric Acid | Total
Number analyzed (Participants) | 16 | 15 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 15 | 31
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 8 | 22
  Male | 2 | 7 | 9
Region of Enrollment [Number; unit: participants]
  United States | 16 | 15 | 31
Body mass index [Mean (Standard Deviation); unit: kg/m2] | 35.9 (3.2) | 38.3 (4.8) | 37.1 (4.1)
Plasma uric acid concentration [Mean (Standard Deviation); unit: mg/dL] | 4.5 (0.2) | 7.1 (1.6) | 5.7 (1.7)

OUTCOME MEASURES:

1. Primary Outcome: Percent Increase in Insulin-stimulated Glucose Uptake
Description: Uric acid will be reduced to 0 with a 30 minute infusion of a uricase (Elitek, Sanofi-Aventis). A hyperinsulinemic-euglycemic clamp procedure in conjunction with stable isotope glucose tracer infusion will be used to measure percent increase in insulin-stimulated glucose uptake in obese subjects with high uric acid before and after uric acid reduction.
Time Frame: 12 hours after reducing uric acid
Measure: Mean (Standard Error); unit: % incr. in insulin-mediated gluc. uptake
Groups:
- Obese Subjects With Normal Uric Acid: Subjects with a body mass index = or > 30 kg/m^2 with normal uric acid (= or < 5 mg/dL)
- Obese Subjects With High Uric Acid: Subjects with a body mass index = or > 30 kg/m^2 with high uric acid (>6 mg/dL)
  Intervention: one single infusion of rasburicase (0.19 mg/kg FFM) infused over 30 min
  Rasburicase: one single infusion of rasburicase (0.19 mg/kg FFM) infused over 30 min
Arm/Group | Obese Subjects With Normal Uric Acid | Obese Subjects With High Uric Acid
Number analyzed (Participants) | 16 | 15
% incr. in insulin-mediated gluc. uptake
  BASAL Insulin Sensitivity | 231 (23) | 162 (24)
  AFTER RASBURICASE Insulin Sensitivity | NA (NA) — Rasburicase infusion to lower uric acid was only administered to subjects in the High Uric Acid group | 156 (17)

2. Secondary Outcome: The Effect of Reducing Uric Acid on Oxidative Status
Description: Uric acid will be reduced to 0 with a 30 minute infusion of a uricase (Elitek, Sanofi-Aventis). Systemic (urinary isoprostanes) and skeletal muscle (carbonylated protein ratio) oxidative stress and total antioxidant capacity (plasma TRAP and FRAP) will be measured in obese subjects with high uric acid before and after uric acid reduction. Levels of isoprostanes were normalized to urinary creatinine and reported at ng/mg.
Time Frame: 12 hours after reducing uric acid
Measure: Mean (Standard Error); unit: ng/mg
Arm/Group | Obese Subjects With Normal Uric Acid | Obese Subjects With High Uric Acid
Number analyzed (Participants) | 16 | 15
ng/mg
  BASELINE urinary isoprostanes | 1.0 (0.15) | 0.68 (0.07)
  AFTER RASBURICASE isoprostanes | NA (NA) — Rasburicase infusion to reduce uric acid was administered only to the High Uric Acid group | 0.96 (0.12)

3. Secondary Outcome: Baseline Carbonylated Protein Ratio
Description: Baseline ratio of total carbonylated proteins to the loading control protein Ran in skeletal muscle
Time Frame: Before reducing uric acid
Measure: Mean (Standard Error); unit: Ratio
Arm/Group | Obese Subjects With Normal Uric Acid | Obese Subjects With High Uric Acid
Number analyzed (Participants) | 16 | 15
Ratio | 929 (86) | 680 (56)

4. Secondary Outcome: AFTER Rasburicase Carbonylated Protein Ratio
Description: Baseline ratio of total carbonylated proteins to the loading control protein Ran in skeletal muscle
Time Frame: 12 hours after reducing uric acid
Population: Analysis only completed on subjects in the High Uric Acid group
Measure: Mean (Standard Error); unit: Ratio
Arm/Group | Obese Subjects With Normal Uric Acid | Obese Subjects With High Uric Acid
Number analyzed (Participants) | 0 | 15
Ratio |  | 1085 (131)

5. Secondary Outcome: Baseline Plasma TRAP
Description: Total Radical-Trapping Antioxidant Potential
Time Frame: Before reducing uric acid
Measure: Mean (Standard Error); unit: mmol · Lˉ¹
Arm/Group | Obese Subjects With Normal Uric Acid | Obese Subjects With High Uric Acid
Number analyzed (Participants) | 16 | 15
mmol · Lˉ¹ | 1.11 (0.02) | 1.31 (0.05)

6. Secondary Outcome: AFTER Rasburicase Plasma TRAP
Description: Total Radical-Trapping Antioxidant Potential
Time Frame: 12 hours after reducing uric acid
Population: AFTER rasburicase plasma Total Radical-Trapping Antioxidant Potential (TRAP) was only measured in the subjects with high uric acid
Measure: Mean (Standard Error); unit: mmol · Lˉ¹
Arm/Group | Obese Subjects With Normal Uric Acid | Obese Subjects With High Uric Acid
Number analyzed (Participants) | 0 | 15
mmol · Lˉ¹ |  | 0.71 (0.02)

7. Secondary Outcome: Baseline Plasma FRAP
Description: Ferric-Reducing Antioxidant Potential
Time Frame: Before reducing uric acid
Measure: Mean (Standard Error); unit: mmol Fe⁺² · Lˉ¹
Groups:
- Obese Subjects With High Uric Acid: Subjects with a body mass index = or > 30 kg/m² with high uric acid (>6 mg/dL)
  Intervention: one single infusion of rasburicase (0.19 mg/kg FFM) infused over 30 min
  Rasburicase: one single infusion of rasburicase (0.19 mg/kg FFM) infused over 30 min
Arm/Group | Obese Subjects With Normal Uric Acid | Obese Subjects With High Uric Acid
Number analyzed (Participants) | 16 | 15
mmol Fe⁺² · Lˉ¹ | 1.03 (0.02) | 1.39 (0.05)

8. Secondary Outcome: AFTER Rasburicase Plasma FRAP (Fe⁺² · Lˉ¹)
Description: Ferric-Reducing Antioxidant Potential
Time Frame: 12 hours after reducing uric acid
Population: AFTER rasburicase plasma FRAP only measured in subjects with high uric acid
Measure: Mean (Standard Error); unit: mmol Fe⁺² · Lˉ¹
Arm/Group | Obese Subjects With Normal Uric Acid | Obese Subjects With High Uric Acid
Number analyzed (Participants) | 0 | 15
mmol Fe⁺² · Lˉ¹ |  | 0.42 (0.02)

ADVERSE EVENTS:
Arm/Group | Obese Subjects With Normal Uric Acid | Obese Subjects With High Uric Acid
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15
Other Adverse Events (participants affected / at risk) | 0/16 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No